CLINICAL TRIAL: NCT03708939
Title: The Role of the Microbiome in Personalized Human Response to Non-caloric Sweeteners
Brief Title: Microbiome and Non-caloric Sweeteners in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weizmann Institute of Science (Other)
Responsible Party: Principal Investigator, Eran Elinav, Prof. Eran Elinav, Weizmann Institute of Science
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 170-2
Record Dates: First submitted 2018-10-14; First posted 2018-10-17 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Glucose Intolerance; Glucose, Low Blood; Glucose, High Blood
MeSH Terms: conditions — Glucose Intolerance | interventions — Glucose; Aspartame; trichlorosucrose; Saccharin; stevioside

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- glucose (Experimental)
  Interventions: Dietary Supplement: Glucose
- aspartame (Experimental)
  Interventions: Dietary Supplement: Aspartame
- sucralose (Experimental)
  Interventions: Dietary Supplement: Sucralose
- saccharin (Experimental)
  Interventions: Dietary Supplement: Saccharin
- Stevia (Experimental)
  Interventions: Dietary Supplement: Stevia
- No supplement control (Experimental)
  Interventions: Other: No Supplement

INTERVENTIONS:
Dietary Supplement: Glucose — Daily consumption of 5g of glucose, for 14 days.
  Arms: glucose
Dietary Supplement: Aspartame — Daily consumption of six commercially available sachets containing aspartame and glucose as bulking agent (1g each sachet), for 14 days.
  Arms: aspartame
Dietary Supplement: Sucralose — Daily consumption of six commercially available sachets containing sucralose and glucose as bulking agent (1g each sachet), for 14 days.
  Arms: sucralose
Dietary Supplement: Saccharin — Daily consumption of six commercially available sachets containing saccharine and glucose as bulking agent (1g each sachet), for 14 days.
  Arms: saccharin
Dietary Supplement: Stevia — Daily consumption of six commercially available sachets containing Stevia and glucose as bulking agent (1g each sachet), for 14 days.
  Arms: Stevia
Other: No Supplement — Follow up without any dietary supplementation.
  Arms: No supplement control

SUMMARY:
Non-caloric sweeteners are common food supplements consumed by millions worldwide as means of combating weight gain and diabetes, by retaining sweet taste without increasing caloric intake. While they are considered safe, there is increasing debate regarding their potential role in contributing to metabolic derangements in some humans. The investigators recently demonstrated that non-caloric sweeteners consumption could induce glucose intolerance in mice and, in preliminary experiments, in distinct human subsets, by functionally altering the gut microbiome, and that the gut microbiome plays an important role in mediating differential glucose responses to identical foods. The proportion of the human population that is susceptible to glucose intolerance induced by non-caloric sweeteners, the common factors that are shared between these individuals and whether and how the microbiome promotes the metabolic derangements remain to be addressed.

ELIGIBILITY:
Inclusion Criteria:

1. BMI<28
2. Age - 18-70
3. Capable of working with smartphone application
4. Capable to work with a glucometer

Exclusion Criteria:

1. Consumption of antibitioics 3 months prior to the first day of the experiment.
2. Consumption of Non caloric sweetners 6 months prior to the first day of the experiment.
3. Diagnosis with type 1 or type 2 diabetes.
4. Pregnancy, fertility treatments
5. Breastfeeding (Including baby to breast and bottle feeding expressed breast milk)
6. Chronic disease (e.g. AIDS, Cushing syndrome, CKD, acromegaly, hyperthyroidism etc.)
7. Cancer and recent anticancer treatment
8. Psychiatric disorders
9. Coagulation disorders
10. IBD (inflammatory bowel diseases)
11. Bariatric surgery
12. Alcohol or substance abuse
13. BMI>28
14. Aspartame group only: phenylketonuria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-02-19 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Blood glucose level | 28 days
  Continuous glucose monitor device

SECONDARY OUTCOMES:
Microbiome | 28 days
  Stool and oral samples

CONTACTS AND LOCATIONS:
Overall Officials: Eran Elinav, Principal Investigator — Weizmann Institute of Science
Locations (1):
- Weizmann Institute of Science, Rehovot, Israel